CLINICAL TRIAL: NCT02747160
Title: Evaluation of an Anxiety Intervention for Older Adults With Cancer and Informal Caregivers of Older Adults With Cancer
Brief Title: Anxiety With Cancer in the Elderly (ACE): A Cognitive-behavioral Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-280
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Anxiety; Depression; Quality of Life
Keywords: Cancer; Anxiety; Cognitive behavior therapy; Elderly; Caregivers
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Managing Anxiety from Cancer (MAC) (Experimental): Older adults with cancer and their primary informal caregiver will receive a six-session cognitive-behavior therapy intervention administered over the telephone by a trained study interventionist. The intervention is administered weekly and each session is 45-50 minutes in length. Patients and caregivers will receive the intervention independently and from separate therapists.
  Interventions: Behavioral: Managing Anxiety from Cancer (MAC)

INTERVENTIONS:
Behavioral: Managing Anxiety from Cancer (MAC) — The intervention consists of six telephone-administered sessions. Session topics include psychoeducation on anxiety, behavioral strategies for managing anxiety, cognitive restructuring, communication skills training, acceptance techniques (patient only), problem-solving strategies (caregiver only), and planning for future anxiety. Session content is tailored for older adults and caregivers of older adults with cancer.

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of and patient adherence to a telephone-administered cognitive-behavioral therapy intervention for anxiety in older adults (65 years and older) with cancer and their primary informal caregiver. This study will also examine whether the intervention has a clinically significant impact on patient anxiety (primary outcome) and depression, distress, and quality of life (secondary outcomes).

DETAILED DESCRIPTION:
This study is a single arm pre-post evaluation of a six-session telephone-administered cognitive-behavioral therapy (CBT) intervention for anxiety in older adults with cancer and their primary informal (unpaid) caregiver. The primary purposes of this study are to evaluate the feasibility of the intervention and study procedures, acceptability of the intervention to older adults with cancer and their primary informal caregiver, and patient and caregiver adherence to the intervention. The secondary purpose is to examine changes in patient and caregiver anxiety, depression, distress, and quality of life pre to post intervention to determine whether the intervention has a clinically significant impact on these outcomes. Anxiety is the primary outcome; depression, distress, and quality of life are secondary outcomes. Patients will be 65 years of age or older and will be recruited from the myeloma, lung, lymphoma, gynecologic, and gastrointestinal cancer clinics at a single institution. Study measures will be administered by telephone prior to initiating the intervention (pre-intervention) and following intervention completion (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 65 years or older
2. Diagnosis of cancer
3. Patient and/or caregiver score of 8 or higher on the anxiety subscale of the Hospital Anxiety and Depression Scale
4. A primary informal caregiver who is willing and able to participate
5. Patient and caregiver are able to communicate over the telephone
6. Caregiver is age 21 years or older.

Exclusion Criteria:

1. Patient or caregiver is not fluent in English
2. Patient or caregiver is too weak or cognitively impaired to participate in the intervention
3. Patient or caregiver has received CBT since the patient's cancer diagnosis
4. Patient or caregiver has an active major psychiatric condition such as schizophrenia
5. Patient only experiences anxiety in the context of a specific medical procedure
6. Patient or caregiver endorses active suicidal ideation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | Post-intervention (6-8 weeks after baseline)
  Attrition rates
Intervention acceptability | Post-intervention (6-8 weeks after baseline)
  Likert scale ratings of perceived helpfulness and readability of the intervention
Patient/caregiver adherence | Post-intervention (6-8 weeks after baseline)
  Sum of number of intervention exercises completed with number of sessions completed by patients and caregivers

SECONDARY OUTCOMES:
Change in anxiety from baseline to post-intervention | Baseline (1-2 weeks after enrollment) and Post-intervention (6-8 weeks after baseline)
  Anxiety sub-scale of the Hospital Anxiety and Depression Scale
Change in distress from baseline to post-intervention | Baseline (1-2 weeks after enrollment) and Post-intervention (6-8 weeks after baseline)
  Distress Thermometer
Emotional health-related quality of life | Baseline (1-2 weeks after enrollment) and Post-intervention (6-8 weeks after baseline)
  Functional Assessment of Cancer Therapy-General: Emotional Quality of Life Sub-Scale; Caregiver Quality of Life-Cancer
Change in depression from baseline to post-intervention | Baseline (1-2 weeks after enrollment) and Post-intervention (6-8 weeks after baseline)
  Depression sub-scale of the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Trevino, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No